CLINICAL TRIAL: NCT02289677
Title: Comparison of the Atmos Scope, the Coopdech and the AirTraq in Pediatric Patients During Resuscitation. Randomized Crossover Manikin Trial
Brief Title: Pediatric Intubation During CPR
Acronym: ETICPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/10
Record Dates: First submitted 2014-11-09; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest
Keywords: intubation; child; resuscitation; simulation; Endotracheal
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intubation during chest compression (Experimental): Intubation during mannequin chest compressions. Chest compression was performed using LUCAS-2 (Physio-Control, Redmond, WA, USA).
  Interventions: Device: ATMOS Scope; Device: COOPDECH; Device: AirTraq

INTERVENTIONS:
Device: ATMOS Scope — Video-laryngoscopy 1
  Other Names: ATMOS Scope Flexible Videoendoscope
Device: COOPDECH — Video-laryngoscopy-1
  Other Names: COOPDECH Video Laryngoscope Portable VLP-100
Device: AirTraq — Optical-laryngoscopy

SUMMARY:
We hypothesized that the video-laryngoscopes are beneficial for intubation of pediatric manikins while performing CPR. In the current study, we compared effectiveness of two video-laryngoscopes (the Coopdech video Laryngoscope portable VLp-100 and the Flexible Videoendoscope: ATMOS Scope) and optical-laryngoscope (the AirTraq) during resuscitation with uninterrupted chest compressions using an child manikin.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medical personnel (physicians, nurses, paramedics)

Exclusion Criteria:

* Not meet the above criteria
* Wrist or Low back diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of first, second and third intubation attempts and overall effectiveness of intubation by participants using two intubation devices

SECONDARY OUTCOMES:
Intubation time | 1 day
  time in seconds required for a successful intubation attempt
POGO score | 1 day
  self-reported percentage of glottis opening (POGO) score
Cormack-Lehane grading | 1 day
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology